CLINICAL TRIAL: NCT05526404
Title: Mobile Application Based Lactulose Titration for Prevention of Hepatic Encephalopathy
Brief Title: Prevention of Hepatic Encephalopathy With Mobile Application Based Lactulose Titration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Douglas (Doug) A. Simonetto, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 22-006646
Record Dates: First submitted 2022-08-31; First posted 2022-09-02 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Hepatic Encephalopathy
MeSH Terms: conditions — Hepatic Encephalopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mobile application-based Bristol stool scale (Experimental): Subjects with cirrhosis who are taking lactulose for the treatment of hepatic encephalopathy will download the Dieta mobile application on their mobile device and take a photo of each bowel movement using the Dieta application
  Interventions: Other: Dieta mobile application

INTERVENTIONS:
Other: Dieta mobile application — Mobile application that functions on mobile phones and allows for tracking of symptoms, dietary intake, and stool characteristics using logs and pictures. Users of the application track symptoms by completing questionnaires regarding stool frequency, consistency, and mental status changes. Users can track dietary intake and stool characteristics by taking time-stamped photos of all dietary intake and bowel movements.

SUMMARY:
This study is being done to assess the safety and efficacy of using mobile application-based Bristol stool scale to titrate lactulose in prevention episodes of hepatic encephalopathy.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written, informed consent.
* Currently taking lactulose daily for prevention of hepatic encephalopathy.

Exclusion Criteria:

* Recent change in dosing of opioid medication.
* Previous Colorectal Surgery.
* Active diarrheal illness.
* Lack of smartphone or other smart device at home.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-09-14 (Actual); Primary Completion 2023-07-08 (Actual); Study Completion 2023-07-08 (Actual)

PRIMARY OUTCOMES:
Achievement of daily stool goal | 4 weeks
  Number of subject to achieve daily stool goal, determined if use of the mobile application leads to improved rates of meeting daily stool goal (3-4 stools per day of Bristol Stool Scale 3-4)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Simonetto, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials